CLINICAL TRIAL: NCT02259309
Title: Immune Modulation by Misoprostol
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Gynuity Health Projects (Other)
Responsible Party: Principal Investigator, David Aronoff, MD, Vanderbilt University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 140667
Record Dates: First submitted 2014-09-22; First posted 2014-10-08 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2016-01

CONDITIONS: Gynecological Infection
Keywords: misoprostol; mucosal; cervical; immune; buccal; vaginal
MeSH Terms: interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Misoprostol administration - buccal then vaginal (Experimental): Vaginal or buccal administration
  Interventions: Drug: Misoprostol - buccal; Drug: Misoprostol - vaginal
- Misoprostol administration - vaginal then buccal (Experimental): Vaginal or buccal administration
  Interventions: Drug: Misoprostol - buccal; Drug: Misoprostol - vaginal

INTERVENTIONS:
Drug: Misoprostol - buccal — buccal administration
  Other Names: Cytotec
Drug: Misoprostol - vaginal — vaginal administration
  Other Names: Cytotec

SUMMARY:
The present study is designed to address the null hypothesis that there is no difference in the local and systemic immunomodulatory effects of buccally or vaginally administered misoprostol in healthy, reproductive-age women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women 18-45 years of age
* Negative result of urine pregnancy test at screening and prior to each administration of study drug
* Normal, regularly occurring menses (being 25-35 day cycles)

Exclusion Criteria:

* Use of hormonal contraception (current or past 3 months)
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) or aspirin within two weeks prior to enrollment or planned use of these medications during the study period
* Allergy to prostaglandins
* Previous cervical cancer
* Partial or complete cervical excision
* Previous hysterectomy
* Immunosuppression: either pharmacological or due to comorbidities
* Diabetes mellitus
* Auto-immune disease
* History of lymphoma or leukemia
* Sexually transmitted infection (by self-report) over previous 1 year
* Bacterial Vaginosis or Candidiasis (current or past 3 months)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparison of misoprostol drug levels in patients after vaginal and buccal administration | Peripheral blood collected at Days 0, 1, 28, and 29
  Peripheral blood collected at Days 0, 1, 28, and 29
Comparison of cytokine and chemokine levels in patients after vaginal and buccal administration | Peripheral blood collected at Days 0, 1, 28, and 29
  Peripheral blood collected at Days 0, 1, 28, and 29
Determination of immune cell activation state after vaginal and buccal administration | Peripheral blood collected at Days 0, 1, 28, and 29
  Peripheral blood collected at Days 0, 1, 28, and 29
Comparison of misoprostol drug levels in patients after vaginal and buccal administration | Cervicovaginal lavage at Days 0, 1, 28, and 29
  Cervicovaginal lavage at Days 0, 1, 28, and 29
Comparison of cytokine and chemokine levels in patients after vaginal and buccal administration | Cervicovaginal lavage at Days 0, 1, 28, and 29
  Cervicovaginal lavage at Days 0, 1, 28, and 29
Determination of immune cell activation state after vaginal and buccal administration | Cervical cytobrush at Days 0, 1, 28, and 29
  Cervical cytobrush at Days 0, 1, 28, and 29

SECONDARY OUTCOMES:
Sequencing of 16S rRNA gene for microbial ecology studies after vaginal and buccal administration | Vaginal swab at Days 0, 1, 28, and 29
  Vaginal swab at Days 0, 1, 28, and 29

CONTACTS AND LOCATIONS:
Overall Officials: David M. Aronoff, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Background] Moran M, Mozes MF, Maddux MS, Veremis S, Bartkus C, Ketel B, Pollak R, Wallemark C, Jonasson O. Prevention of acute graft rejection by the prostaglandin E1 analogue misoprostol in renal-transplant recipients treated with cyclosporine and prednisone. N Engl J Med. 1990 Apr 26;322(17):1183-8. doi: 10.1056/NEJM199004263221703. PMID 2109195
- [Background] Pouteil-Noble C, Chapuis F, Berra N, Hadj-Aissa A, Lacavalerie B, Lefrancois N, Martin X, Touraine JL. Misoprostol in renal transplant recipients: a prospective, randomized, controlled study on the prevention of acute rejection episodes and cyclosporin A nephrotoxicity. Nephrol Dial Transplant. 1994;9(5):552-5. doi: 10.1093/ndt/9.5.552. PMID 8090337
- [Background] Zieman M, Fong SK, Benowitz NL, Banskter D, Darney PD. Absorption kinetics of misoprostol with oral or vaginal administration. Obstet Gynecol. 1997 Jul;90(1):88-92. doi: 10.1016/S0029-7844(97)00111-7. PMID 9207820
- [Background] Waiser J, Bohler T, Stoll J, Schumann B, Budde K, Neumayer HH. The immunosuppressive potential of misoprostol--efficacy and variability. Clin Immunol. 2003 Dec;109(3):288-94. doi: 10.1016/j.clim.2003.08.009. PMID 14697743
- [Background] Middleton T, Schaff E, Fielding SL, Scahill M, Shannon C, Westheimer E, Wilkinson T, Winikoff B. Randomized trial of mifepristone and buccal or vaginal misoprostol for abortion through 56 days of last menstrual period. Contraception. 2005 Nov;72(5):328-32. doi: 10.1016/j.contraception.2005.05.017. Epub 2005 Aug 9. PMID 16246656
- [Background] Tang OS, Ho PC. The pharmacokinetics and different regimens of misoprostol in early first-trimester medical abortion. Contraception. 2006 Jul;74(1):26-30. doi: 10.1016/j.contraception.2006.03.005. Epub 2006 Apr 27. PMID 16781256
- [Background] el-Refaey H, Rajasekar D, Abdalla M, Calder L, Templeton A. Induction of abortion with mifepristone (RU 486) and oral or vaginal misoprostol. N Engl J Med. 1995 Apr 13;332(15):983-7. doi: 10.1056/NEJM199504133321502. PMID 7885426
- [Background] Ho PC, Ngai SW, Liu KL, Wong GC, Lee SW. Vaginal misoprostol compared with oral misoprostol in termination of second-trimester pregnancy. Obstet Gynecol. 1997 Nov;90(5):735-8. doi: 10.1016/S0029-7844(97)00419-5. PMID 9351755
- [Background] Silverstein FE, Graham DY, Senior JR, Davies HW, Struthers BJ, Bittman RM, Geis GS. Misoprostol reduces serious gastrointestinal complications in patients with rheumatoid arthritis receiving nonsteroidal anti-inflammatory drugs. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 1995 Aug 15;123(4):241-9. doi: 10.7326/0003-4819-123-4-199508150-00001. PMID 7611589
- [Background] Herting RL, Clay GA. Overview of clinical safety with misoprostol. Dig Dis Sci. 1985 Nov;30(11 Suppl):185S-193S. doi: 10.1007/BF01309407. PMID 3932053
- [Background] Wildeman RA. Focus on misoprostol: review of worldwide safety data. Clin Invest Med. 1987 May;10(3):243-5. PMID 3113801
- [Background] Rostom A, Dube C, Wells G, Tugwell P, Welch V, Jolicoeur E, McGowan J. Prevention of NSAID-induced gastroduodenal ulcers. Cochrane Database Syst Rev. 2002;(4):CD002296. doi: 10.1002/14651858.CD002296. PMID 12519573
- [Background] Chong E, Tsereteli T, Nguyen NN, Winikoff B. A randomized controlled trial of different buccal misoprostol doses in mifepristone medical abortion. Contraception. 2012 Sep;86(3):251-6. doi: 10.1016/j.contraception.2011.12.012. Epub 2012 Feb 2. PMID 22305917
- [Background] Raymond EG, Shannon C, Weaver MA, Winikoff B. First-trimester medical abortion with mifepristone 200 mg and misoprostol: a systematic review. Contraception. 2013 Jan;87(1):26-37. doi: 10.1016/j.contraception.2012.06.011. Epub 2012 Aug 13. PMID 22898359
- [Background] Kotsonis FN, Dodd DC, Regnier B, Kohn FE. Preclinical toxicology profile of misoprostol. Dig Dis Sci. 1985 Nov;30(11 Suppl):142S-146S. doi: 10.1007/BF01309401. PMID 3932047
- [Background] Zane S, Guarner J. Gynecologic clostridial toxic shock in women of reproductive age. Curr Infect Dis Rep. 2011 Dec;13(6):561-70. doi: 10.1007/s11908-011-0207-7. PMID 21882086
- [Background] Fjerstad M, Trussell J, Sivin I, Lichtenberg ES, Cullins V. Rates of serious infection after changes in regimens for medical abortion. N Engl J Med. 2009 Jul 9;361(2):145-51. doi: 10.1056/NEJMoa0809146. PMID 19587339
- [Background] Hemmerling A. The safety of misoprostol. ELSEVIER IRELAND LTD; 2006.